CLINICAL TRIAL: NCT02919176
Title: The Activation of Brown and Beige Fat and Role in Insulin Sensitivity
Brief Title: Brown Fat Activation Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-0642-F1V; R01DK112282 (NIH)
Record Dates: First submitted 2016-08-22; First posted 2016-09-29 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Obese; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — mirabegron; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Mirabegron (Active Comparator): Mirabegron 50 mg/day
  Interventions: Drug: Mirabegron
- Pioglitazone (Active Comparator): Pioglitazone 30 mg/day
  Interventions: Drug: Pioglitazone
- Mirabegron and Pioglitazone (Experimental): Combination of Mirabegron 50 mg/day and Pioglitazone 30 mg/day
  Interventions: Drug: Mirabegron and Pioglitazone

INTERVENTIONS:
Drug: Mirabegron — Mirabegron 50 mg/day
  Other Names: MYRBETRIQ
  Arms: Mirabegron
Drug: Pioglitazone — Pioglitazone 30 mg/day
  Other Names: ACTOS
  Arms: Pioglitazone
Drug: Mirabegron and Pioglitazone — Mirabegron 50 mg/day and Pioglitazone 30 mg/day
  Other Names: MYRBETRIQ and ACTOS
  Arms: Mirabegron and Pioglitazone

SUMMARY:
This is an open lable, pilot study in which the investigator will research the effect of two FDA approved drugs, Mirabegron and Pioglitazone on fat tissue.

Pioglitazone is drug approved by the FDA for the treatment of diabetes and Mirabegron is a drug that is approved by the FDA for the treatment of overactive bladder. These drugs are not approved by the FDA for the purposes being studied in this research. Therefore, the way in which the investigator intends to use them in this study are considered investigational.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the amount and activity of brown adipose tissue (BAT) and beige adipose can be increased with the use of Mirabegron or Pioglitazone, alone or in combination.

The research procedures will be conducted at the University of Kentucky (UK) Medical Center at the Center for Clinical Translational Sciences research unit (CCTS). Study participants will need to come to the CCTS Unit for approximately 9 visits, as outlined below. Most of these visits will be less than 1 hour, but 3 visit will involve procedures and will vary in time ranging from 4 hour to 8 hours. Thus, a participant's total participation will be approximately 9 visits over the next 12 weeks.

After passing the screening phase, participants will be randomized (like the flipping of coin) at Visit 4 to one of three treatment groups and the participant will stay in their assigned treatment group during their entire participation in the study. The three groups are:

* Group M: Mirabegron 50 mg/day
* Group P: Pioglitazone 30 mg/day
* Group MP: combination Mirabegron 50 mg/day and Pioglitazone 30 mg/day

Fasting requirements: Nothing to eat after 9 pm the night before a specific test or procedure.

Glucose tolerance test and fasting lab tests: This will be a standard oral glucose tolerance test using 75 g of glucose, with blood for glucose and insulin drawn at times 0, 30, 60, 90, and 120 min. This test will determine if the participants have impaired glucose tolerance, diabetes, or are normal. This fasting blood sample will be used to conduct routine blood tests that are a normal part of a physical exam, such as cholesterol, liver enzymes and electrolytes.

Based on the blood tests, the oral glucose tolerance test (OGTT), and other measurements, the investigator will determine whether a participant has impaired glucose tolerance or a normal glucose level, and whether they fit the other criteria of the study.

Body Mass Index and DXA Scan: The investigator will record the participant's weight, height, waist and hip measurements. Measurement of total body fat will be performed to determine the participant's percent body fat using dual energy X-ray absorptiometry (DXA). DXA uses very low levels of X-ray to measure the amount of fat, muscle, and bone in different body areas. Participants will be asked to lie on a table while wearing light clothing or a gown.

Positron Emission Tomography (PET) Scan: A PET scan is a type of imaging test. It uses a radioactive substance called a tracer to look for high areas of metabolic activity in the body. A PET scan is a standard test performed for certain conditions, and in this instance it is being used to see a participant's brown fat. 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) is an FDA-approved drug that is injected into the body before a PET scan, and used as a "tracer" to help light up the areas the doctors need to see. The investigators is not studying the effectiveness of this drug in this study.

To see the brown fat, the investigator will first need to make a participant cold. To do this, a participant will change into loose fitting light clothing, and then place around their midsection, a special jacket, and cold water will circulate through this jacket for 1 hr.

The jacket is then removed, and the participants are injected through a vein (IV) with the FDG tracer. The IV needle is most often inserted on the inside of the elbow. The tracer travels through the blood and collects in organs and tissues. This helps the radiologist see certain areas more clearly.

Participants will lie on a narrow table that slides into a large tunnel-shaped scanner. The PET detects signals from the tracer. A computer changes the signals into 3D pictures. The images are displayed on a monitor for the radiologist to read.

Fat biopsies: After an overnight fast, the biopsy procedures will be performed as follows: A fat sample (called a fat biopsy) will be removed by the investigator from the lower abdomen and from the thigh. The skin at the biopsy sites will be anesthetized using the local anesthetic, lidocaine, then a 1 incision will be made on the abdomen and a ½ inch incision on thigh, through the skin, and a small amount of fat tissue will be removed. The incisions will then be closed using stitches. Participants will have a total of 4 fat biopsies: Two prior to receiving study drug (at any time between visits 2-4) and two while taking the study drug (at any time between visits 6-9).

Muscle biopsy. At the time of the thigh adipose biopsy, a muscle biopsy is performed through the same skin incision. Participants will have a total of 2 muscle biopsies: 1 prior to receiving study drug (at any time between visits 2-4) and one while taking the study drug (at any time between visits 6-9).

Euglycemic clamp: Insulin sensitivity will be measured using a clamp. Participants will come to the CCTS after fasting overnight. Two intravenous plastic tubes will be inserted into veins in their arm. Participants will then be given a constant injection of glucose along with a constant injection of insulin. The glucose and insulin are balanced such that the participant's blood glucose stays constant between about 90-100 mg/dl. Blood will then be drawn from the intravenous line frequently (about every 5-10 minutes) for measurement of blood glucose and insulin. These blood measurements will continue for 4 hours; the total amount of blood that will be withdrawn will be about 100 cc (about 6 tablespoons), which is about one quarter as much as would be taken if the participant were to donate blood.

Urine Collection: Females who are capable of getting pregnant, will also be asked to give a sample of urine to test for pregnancy. If the test results positive for pregnancy, participants will not be able to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* slightly abnormal blood sugar (A1C between 5.7 and 6.5 or impaired glucose tolerance)
* Metabolic Syndrome features (hypertension, abnormal lipids, abdominal obesity)
* Body Mass Index between 27-45
* Ambulatory

Exclusion Criteria:

* A history of heart disease
* Cancer or a history of cancer within the last 5 years
* Kidney disease
* Currently taking steroids or anticoagulants
* A chronic inflammatory condition such as rheumatoid arthritis or inflammatory bowel disease
* A body mass index (BMI) greater than 45
* Diabetes or the chronic use of any antidiabetic medications
* Uncontrolled blood pressure, urinary retention, overactive thyroid
* Significant swelling in hands, feet, face, arms.
* Currently taking β-blockers
* Daily use of NSAIDS or other anti-inflammatory drugs (eg. corticosteroids)
* Using low-dose aspirin (Participants will need to discontinue use for 7 days prior to the biopsies)
* Antiplatelet medication or blood thinners (examples: Aspirin, warfarin, Effient, Plavix)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Change in beige adipose tissue | baseline and after 10 weeks of treatment
  Beige adipose tissue markers will be evaluated at baseline, and after treatment with mirabegron, pioglitazone, or both drugs
Change in brown adipose tissue | baseline and after 10 weeks of treatment
  Brown adipose tissue will be evaluated by PET-CT scan at baseline, and after treatment with mirabegron, pioglitazone, or both drugs
Change in insulin sensitivity | baseline and after 10 weeks of treatment
  Insulin sensitivity will be assessed at baseline and after treatment with mirabegron, pioglitazone, or both drugs, using a euglycemic clamp

SECONDARY OUTCOMES:
Change in body mass index | baseline and after 10 weeks of treatment
  Body mass index will be assessed at baseline and after treatment with mirabegron, pioglitazone, or both drugs
Change in glucose tolerance | baseline and after 10 weeks of treatment
  Using an oral glucose tolerance test, glucose tolerance will be assessed at baseline and after treatment with mirabegron, pioglitazone, or both drugs

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, MD, Principal Investigator — University of Kentucky
Locations (1):
- Center for Clinical and Translational Science, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finlin BS, Memetimin H, Zhu B, Confides AL, Vekaria HJ, El Khouli RH, Johnson ZR, Westgate PM, Chen J, Morris AJ, Sullivan PG, Dupont-Versteegden EE, Kern PA. The beta3-adrenergic receptor agonist mirabegron improves glucose homeostasis in obese humans. J Clin Invest. 2020 May 1;130(5):2319-2331. doi: 10.1172/JCI134892. PMID 31961829
- [Derived] Finlin BS, Memetimin H, Zhu B, Confides AL, Vekaria HJ, El Khouli RH, Johnson ZR, Westgate PM, Chen J, Morris AJ, Sullivan PG, Dupont-Versteegden EE, Kern PA. Pioglitazone does not synergize with mirabegron to increase beige fat or further improve glucose metabolism. JCI Insight. 2021 Mar 22;6(6):e143650. doi: 10.1172/jci.insight.143650. PMID 33571166
- [Derived] Finlin BS, Memetimin H, Confides AL, Kasza I, Zhu B, Vekaria HJ, Harfmann B, Jones KA, Johnson ZR, Westgate PM, Alexander CM, Sullivan PG, Dupont-Versteegden EE, Kern PA. Human adipose beiging in response to cold and mirabegron. JCI Insight. 2018 Aug 9;3(15):e121510. doi: 10.1172/jci.insight.121510. eCollection 2018 Aug 9. PMID 30089732

DOCUMENTS (1):
  • Informed Consent Form (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT02919176/ICF_000.pdf